CLINICAL TRIAL: NCT01144689
Title: Assessing Mindfulness Training as a Mechanistic Probe for Stress-Induced Brain Activation and Relapse Prevention for Tobacco Addiction
Brief Title: Mindfulness Training for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0808004113
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Cigarette Smoking; Tobacco Smoking; Nicotine Dependence; Smoking Cessation
Keywords: mindfulness; smoking; stress
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder; Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Training (Experimental)
  Interventions: Behavioral: Mindfulness Training
- Smoking Cessation Therapy (Active Comparator)
  Interventions: Behavioral: Smoking Cessation Therapy

INTERVENTIONS:
Behavioral: Mindfulness Training — 8 sessions of behavioral treatment for smoking cessation
  Arms: Mindfulness Training
Behavioral: Smoking Cessation Therapy — 8 sessions of behavioral treatment for smoking cessation
  Arms: Smoking Cessation Therapy

SUMMARY:
The purpose of this study is to assess the effects of mindfulness training (MT) compared to standard Smoking Cessation Therapy (SCT) on smoking cessation and stress provocation in individuals trying to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 60
2. Smoking 10 or more cigarettes per day
3. Fewer than 3 months of smoking abstinence in the past year
4. Motivated to stop smoking

Exclusion Criteria:

1. Current use of psychoactive medications that have not been at a stable dose for the past six months, are used as mood stabilizers, or are used as smoking cessation treatments. Individuals who are on psychoactive medications that are stable, not mood stabilizers, and not used for smoking cessations are excluded from fMRI sessions but not smoking cessation treatment.
2. Use of another investigational drug within 30 days
3. Any serious or unstable disease within 6 months
4. Meets criteria for substance dependence within the past year
5. Left handed (will be excluded from fMRI only)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Between group differences in continuous abstinence | during treatment and 6, 12 and 18 weeks after treatment initiation

SECONDARY OUTCOMES:
Between group differences in perceived stress | 6, 12 and 18 weeks after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Brewer JA, Mallik S, Babuscio TA, Nich C, Johnson HE, Deleone CM, Minnix-Cotton CA, Byrne SA, Kober H, Weinstein AJ, Carroll KM, Rounsaville BJ. Mindfulness training for smoking cessation: results from a randomized controlled trial. Drug Alcohol Depend. 2011 Dec 1;119(1-2):72-80. doi: 10.1016/j.drugalcdep.2011.05.027. Epub 2011 Jul 1. PMID 21723049
- [Result] Elwafi HM, Witkiewitz K, Mallik S, Thornhill TA 4th, Brewer JA. Mindfulness training for smoking cessation: moderation of the relationship between craving and cigarette use. Drug Alcohol Depend. 2013 Jun 1;130(1-3):222-9. doi: 10.1016/j.drugalcdep.2012.11.015. Epub 2012 Dec 21. PMID 23265088
- [Derived] Kober H, Brewer JA, Height KL, Sinha R. Neural stress reactivity relates to smoking outcomes and differentiates between mindfulness and cognitive-behavioral treatments. Neuroimage. 2017 May 1;151:4-13. doi: 10.1016/j.neuroimage.2016.09.042. Epub 2016 Sep 28. PMID 27693614